CLINICAL TRIAL: NCT03046017
Title: Neuromodulation of Lidocaine Cream Effect on Chronic Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015P001440
Record Dates: First submitted 2017-01-27; First posted 2017-02-08 (Estimated); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- real tDCS (Active Comparator): In this group, the tDCS stimulates areas of the brain being examined in this study to increase their activity.
  Interventions: Device: tDCS; Other: Lidocaine cream; Other: Control cream
- sham tDCS (Sham Comparator): In this group, sham tDCS does not provide real stimulation though participants will not know this until the debriefing at the end of the study. Sham will be used to determine if the results of this study are due to the tDCS or other reasons.
  Interventions: Device: tDCS; Other: Lidocaine cream; Other: Control cream
- control group (Other): In this group, participants will receive tDCS but will only receive a cream on their lower back.
  Interventions: Device: tDCS; Other: Lidocaine cream; Other: Control cream

INTERVENTIONS:
Device: tDCS — Electrical stimulation will be applied on the head to temporarily influence brain activity in specific regions.
Other: Lidocaine cream — Lidocaine cream will be applied to reduce pain sensitivity (analgesia).
Other: Control cream — A neutral cream will be applied as a control.

SUMMARY:
Chronic low back pain patients aged 21 to 60 needed for a research study of the effects of transcranial direct current stimulation (tDCS) on the analgesic effects of lidocaine cream as measured by functional Magnetic Resonance Imaging (fMRI). Study will be conducted on nine separate days not requiring an overnight stay in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers 21-60 years of age.
* Meets the Classification Criteria of chronic LBP (having low back pain for more than 6 months), as determined by the referring physician.
* At least 4/10 clinical pain on the 11-point LBP VAS (criteria recommended by Dworkin et al.)
* At least a 10th grade English-reading level; English can be a second language provided that the patients understand all questions used in the assessment measures.

Exclusion Criteria:

* Specific causes of back pain (e.g., cancer, fractures, spinal stenosis, infections).
* Complicated back problems (e.g., prior back surgery, medicolegal issues).
* The intent to undergo surgery during the time of involvement in the study.
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma, claustrophobia, epilepsy or acute eczema under the electrodes.
* Presence of any contraindications to MRI scanning. For example: cardiac pacemaker, metal implants, claustrophobia, pregnancy, cannot lie still in an fMRI scanner.
* History of medical or psychiatric illness.
* History of substance / alcohol abuse or dependence.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
fMRI signal changes | 2 days; Sessions 5 and 7
Gracely Scale pain rating changes | 2 days; Sessions 2 and 7
resting state functional connectivity changes | 2 days; Sessions 5 and 7

CONTACTS AND LOCATIONS:
Locations (1):
- Martinos Center for Biomedical Imagin, Charlestown, Massachusetts, United States